CLINICAL TRIAL: NCT02080494
Title: Tranexamic Acid in Orthopaedic Trauma Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-036
Record Dates: First submitted 2014-01-08; First posted 2014-03-06 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-05

CONDITIONS: Blood Loss; Trauma; Fracture; Surgery
Keywords: tranexamic acid; orthopaedic trauma; pelvic fracture; hip fracture; femur fracture; blood loss
MeSH Terms: conditions — Hemorrhage; Wounds and Injuries; Fractures, Bone; Hip Fractures; Femoral Fractures | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No tranexamic acid given
- Tranexamic Acid (Experimental): 15 mg/kg preoperative IV dose followed by another 15 mg/kg IV dose three hours after the initial dose
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid

SUMMARY:
Tranexamic acid is an antifibrinolytic drug that has been used to decrease post-operative blood loss. This study is a prospective, randomized controlled trial investigating the use of tranexamic acid in fracture surgery around the hip and knee, in which significant blood loss (>300mL) is expected.

The hypothesis of this study is that tranexamic acid will be associated with a decrease in post-operative blood loss, as well as a decreased need for allogenic blood transfusion, in patients who have fracture surgery around the hip and knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated fractures of the pelvic ring, acetabulum, femur or tibia that will require open reduction and internal fixation
* Expected blood loss is greater than 300 mL
* Age ≥ 18
* Skeletal maturity

Exclusion Criteria:

* Pregnant or breastfeeding
* Patients taking oral contraceptives
* Contraindication to venous thromboembolic event (VTE) prophylaxis (intracranial, intrathoracic, intra-abdominal bleeding or spine fractures)
* Patients requiring operative intervention for other injuries (orthopaedic or non-orthopaedic)
* Known hypercoagulable state including history of prescribed anti-coagulation (warfarin, plavix, low molecular weight heparin)
* Renal Insufficiency (creatinine greater than 1.5mg/dL)
* Open fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-05; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
hemoglobin value | through postoperative day four

SECONDARY OUTCOMES:
hematocrit value | through postoperative day four
number of units of allogenic blood transfused | through postoperative day four

CONTACTS AND LOCATIONS:
Overall Officials: Dirk W Kiner, MD, Principal Investigator — UTCOM Chattanooga / Erlanger Health System
Locations (1):
- Erlanger Health System, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No